CLINICAL TRIAL: NCT00450372
Title: Clinical Protocol for Phase II Testing of ADI-PEG 20 in Patients With Metastatic Melanoma
Brief Title: Pegylated Arginine Deiminase in Treating Patients With Metastatic Melanoma That Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20030698; SCCC-2003045
Record Dates: First submitted 2007-03-20; First posted 2007-03-22 (Estimated); Results first posted 2013-05-01 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2016-12

CONDITIONS: Melanoma (Skin)
Keywords: recurrent melanoma; stage IV melanoma
MeSH Terms: conditions — Melanoma | interventions — ADI PEG20; arginine deiminase; Polyethylene Glycols

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ADI-PEG 20 (Experimental)
  Interventions: Biological: ADI-PEG-20; Other: Pharmacology Studies

INTERVENTIONS:
Biological: ADI-PEG-20 — There will be 6 cycles planned, each consisting of 4 weeks. During each cycle subjects will receive injections on days 1, 8, 15, and 22 + 2 days. All subjects may begin treatment with 160 IU/m2 on a weekly basis.
  Other Names: Arginine Deiminase (ADI) formulated with polyethylene glycol (PEG)
Other: Pharmacology Studies — tissue blocks will be obtained from the initial biopsy of melanoma. Immunohistochemical staining for ASS and RT-PCR will be performed on the tumor tissue

SUMMARY:
RATIONALE: Pegylated arginine deiminase may stop the growth of tumor cells by taking away an amino acid needed for cell growth.

PURPOSE: This phase II trial is studying how well pegylated arginine deiminase works in treating patients with metastatic melanoma that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary:

* Determine the clinical response (complete and partial response) in patients with unresectable metastatic melanoma treated with pegylated arginine deiminase.

Secondary:

* Determine the toxicity profile of this drug in these patients.
* Determine the pharmacokinetics and pharmacodynamics of this drug in these patients.
* Determine the progression-free survival and overall survival of patients treated with this drug.

OUTLINE: Patients receive pegylated arginine deiminase intramuscularly once or twice a week in weeks 1-4. Courses repeat every 4 weeks for 6 courses in the absence of disease progression or unacceptable toxicity.

Blood samples are acquired at baseline and every 2 weeks thereafter for pharmacokinetic and pharmacodynamic studies.

After completion of study treatment, patients are followed every 3 months for 1 year, every 6 months for 5 years, and annually thereafter.

PROJECTED ACCRUAL: A total of 43 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic melanoma, meeting any of the following criteria:

  * Progressive disease after chemotherapy, radiotherapy, surgery, or immunotherapy
  * No longer responding to standard therapy OR have refused standard therapy
* Unresectable disease
* Measurable or evaluable disease
* No clinical ascites
* No symptomatic pleural effusion

PATIENT CHARACTERISTICS:

* Life expectancy ≥ 12 weeks
* Karnofsky performance status 70-100%
* Bilirubin ≤ 3.0 mg/dL
* Albumin ≥ 3.0 g/dL
* Alkaline phosphatase < 5 times upper limit of normal (ULN)
* Serum glucose > 60 mg/dL
* Amylase < 1.5 times ULN
* Absolute neutrophil count > 1,500/mm³
* Platelet count > 100,000/mm³
* No New York Heart Association class III-IV heart failure
* No serious infection requiring treatment with antibiotics
* No known allergy to E. coli drug products (e.g., sargramostim [GM-CSF])
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use 2 forms of effective contraception

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 4 weeks since prior anticancer therapy
* At least 4 weeks since prior surgery and recovered
* No concurrent participation in another investigational drug study

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2004-06; Primary Completion 2011-01 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynn G. Feun, MD, Study Chair — University of Miami Sylvester Comprehensive Cancer Center
Locations (1):
- University of Miami Sylvester Comprehensive Cancer Center - Miami, Miami, Florida, United States

REFERENCES:
- [Result] Feun LG, Marini A, Walker G, Elgart G, Moffat F, Rodgers SE, Wu CJ, You M, Wangpaichitr M, Kuo MT, Sisson W, Jungbluth AA, Bomalaski J, Savaraj N. Negative argininosuccinate synthetase expression in melanoma tumours may predict clinical benefit from arginine-depleting therapy with pegylated arginine deiminase. Br J Cancer. 2012 Apr 24;106(9):1481-5. doi: 10.1038/bjc.2012.106. PMID 22472884

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Arm
Started | 38
Completed | 37
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm
Number analyzed (Participants) | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 25
Age, Continuous [Mean (Full Range); unit: years] | 69 [25 to 85]
Gender [Count of Participants; unit: Participants]
  Female | 13
  Male | 25
Region of Enrollment [Number; unit: participants]
  United States | 38

OUTCOME MEASURES:

1. Primary Outcome: Response Rate (Partial and Complete Response) in Patients With or Without ASS Expression Present in Tumor.
Description: Response rate is defined as a partial response, PR, and complete response, CR, lasting for at least 30 days per RECIST criteria, v. 1.0. Complete response will be defined as disappearance of all target lesions. Partial response will be defined as at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference the baseline sum of LD
Time Frame: Up to 16 months
Population: Of the 38 subjects enrolled, only 10 were ASS-positive and 17 were ASS-negative. The remaining 11 subjects, who declined pre-treatment biopsies, were not assessed.
Measure: Number; unit: participants
Groups:
- ADI-PED 20: Argininosuccinate Synthetase Positive (ASS+): Patients with Argininosuccinate Synthetase (ASS) expression present in tumor
- ADI-PEG 20: Argininosuccinate Synthetase Negative (ASS-): Patients without Argininosuccinate Synthetase (ASS) expression present in tumor
Arm/Group | ADI-PED 20: Argininosuccinate Synthetase Positive (ASS+) | ADI-PEG 20: Argininosuccinate Synthetase Negative (ASS-)
Number analyzed (Participants) | 10 | 17
participants | 0 | 4

2. Secondary Outcome: Median Overall Survival
Description: Overall survival will be estimated using the product-limit method of Kaplan & Meier.
Time Frame: Up to 16 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Groups:
- ADI-PEG 20: Argininosuccinate Synthetase Positive (ASS+): Patients with ASS expression present in tumor
- ADI-PEG 20: Argininosuccinate Synthetase Negative (ASS-): Patients without ASS expression in tumor
Arm/Group | ADI-PEG 20: Argininosuccinate Synthetase Positive (ASS+) | ADI-PEG 20: Argininosuccinate Synthetase Negative (ASS-)
Number analyzed (Participants) | 10 | 17
months | 9.3 [2.5 to 9.3] | 14.6 [4.4 to 14.6]

3. Secondary Outcome: Median Time to Progression
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: Up to 16 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | ADI-PEG 20: Argininosuccinate Synthetase Positive (ASS+) | ADI-PEG 20: Argininosuccinate Synthetase Negative (ASS-)
Number analyzed (Participants) | 10 | 17
months | 1.8 [0.7 to 3.4] | 3.6 [1.6 to 12.7]

ADVERSE EVENTS:
Arm/Group | Single Arm
Serious Adverse Events (participants affected / at risk) | 9/37
Other Adverse Events (participants affected / at risk) | 5/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm (N=37)
Allergic Reaction (Injury, poisoning and procedural complications) | 1 — Grade 3
Neutropenia - Grade 3 (Blood and lymphatic system disorders) | 3 — Grade 3
Neutropenia - Grade 4 (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 — Grade 4
Anaemia (Blood and lymphatic system disorders) | 1 — Grade 3
Fatigue (General disorders) | 2 — Grade 3
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm (N=37)
Myelosuppression (Blood and lymphatic system disorders) | 5

LIMITATIONS AND CAVEATS:
Of the 38 subjects enrolled, only 10 were ASS-positive and 17 were ASS-negative. The remaining 11 subjects, who declined pre-treatment biopsies, were not assessed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes